CLINICAL TRIAL: NCT05490030
Title: A Phase 1, Open-label, Single-dose, Multi-center, Parallel Group Study to Evaluate the Pharmacokinetics of TNO155 in Participants With Mild, Moderate, or Severe Hepatic Impairment Compared to Matched Healthy Control Participants
Brief Title: Pharmacokinetics of TNO155 in Participants With Mild, Moderate, or Severe Hepatic Impairment Compared to Matched Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTNO155A12106
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hepatic Impairment
Keywords: Hepatic; Impairment; TNO155; Phase 1; pharmacokinetics; safety; Tolerability; Child-Pug

STUDY DESIGN:
Intervention Model Description: The study will be divided into 2 parts. Participants in the hepatic impairment groups will be staged by their respective degree of hepatic impairment according to the Child Pugh classification score determined at the screening visit and confirmed unchanged at the baseline visit.
  Healthy participants who were identified and enrolled as matching partners for a hepatic impairment group in Part I can serve as matching partners for participants in hepatic impairment group in Part II if they fulfilled the matching criteria. Otherwise, additional matched healthy participants will be enrolled.
  Part I: will include participants with mild and moderate levels of hepatic impairment as well as healthy control participants assigned to the groups Part II: will include participants with severe hepatic impairment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (control) (Experimental): Healthy control participants with normal hepatic function
  Interventions: Drug: TNO155
- Group 2 (score 5-6) (Experimental): Mild hepatic impairment: Child-Pugh A
  Interventions: Drug: TNO155
- Group 3 (score 7-9) (Experimental): Moderate hepatic impairment: Child-Pugh B
  Interventions: Drug: TNO155
- Group 4 (score 10-15) (Experimental): Severe hepatic impairment: Child-Pugh C. This group may be opened if allowed by the results of the interim analysis of the Groups 1 to 3.
  Interventions: Drug: TNO155

INTERVENTIONS:
Drug: TNO155 — Single oral dose of TNO155 on Day 1

SUMMARY:
The purpose of this study is to evaluate the effect of various degrees of hepatic impairment on plasma pharmacokinetics (PK), safety and tolerability of TNO155.

The results of this study will guide the Novartis recommendation regarding whether or not a dose adjustment may be needed when treating patients with hepatic impairment.

DETAILED DESCRIPTION:
This is a study to evaluate the PK of TNO155 in participants with mild, moderate or severe hepatic impairment compared to matched healthy control participants with normal hepatic function.

The study will be divided into 2 parts. Participants in the hepatic impairment groups will be staged by their respective degree of hepatic impairment (mild, moderate, or severe) according to a classification score determined at the screening visit and confirmed unchanged at the baseline visit.

Each participant in the healthy control group may be matched to 1 or more evaluable participants with hepatic impairment with respect to age (± 10 years), body weight (± 20%), sex and smoking status (smoker vs. non smoker). Each participant in the control group can be matched to participants from any hepatic impairment group but cannot be matched to more than 1 participant from the same hepatic impairment group.

All participants will be domiciled from Day -1 until Day 11. All participants should have a poststudy safety follow-up contact conducted approximately 30 days after administration of study treatment. The study will be considered complete once all the participants have finished the required assessments, dropped out, or been lost to follow-up before completing the required assessments.

ELIGIBILITY:
Inclusion Criteria:

All participants Participants must weigh at least 50 kg and no more than 120 kg and must have a body mass index (BMI) within the range of 18.0 to 38.0 kg/m2, inclusive, for healthy participants. For participants with hepatic impairment without overt ascites, the BMI should be within the range of 18.0 to 40.0 kg/m2. For participants with hepatic impairment with overt ascites, the BMI should be within the range of 18.0 to 45.0 kg/m2.

Group 1

•Each healthy control participant must match in age (± 10 years), sex, body weight (± 20%), and smoking status to at least 1 hepatic impairment participant in Groups 2, 3 and/or 4.

Groups 2 to 4 •Participants with mild, moderate or severe hepatic impairment must have a Child-Pugh score clinically determined at screening and confirmed unchanged at baseline calculated as per the Child-Pugh classification in line with the hepatic impairment status of each Group

Exclusion Criteria:

All Participants

* Use of drugs (prescription, non-prescription and herbal remedies such as St John's wort) known to affect CYP3A or UGT1A3, including UGT1A3 inhibitors and inducers and strong and moderate CYP3A inhibitors and inducers, within 4 weeks prior to dosing until completion of the End of Study Visit.
* Acute or chronic hepatitis B or C infection or active infection requiring therapy that will not be completed before screening.

Left ventricular ejection fraction (LVEF) < 50% or below the institutional standard lower limit, whichever is higher, as determined by multiple gated acquisition (MUGA) scan or Trans-thoracic echocardiography (TTE) at screening or baseline.

•At screening, history of retinal vein occlusion (RVO) or presence of predisposing factors to RVO or central serous retinopathy, or any other clinically significant ophthalmologic abnormalities determined by an ophthalmologist.

Group 1

* Any single parameter of alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT), or alkaline phosphatase (ALP) exceeding 2.5 × upper limit of normal (ULN) or total bilirubin ≥ 1.5 ULN OR any elevation above ULN of more than 1 parameter of ALT, AST, GGT, ALP, or serum bilirubin at screening or baseline.
* Impaired renal function as indicated by clinically significantly abnormal creatinine or blood urea nitrogen and/or other urea values outside local laboratory ranges or abnormal urinary constituents at screening or baseline.

Groups 2 and 3

* Severe complications of liver disease within the preceding 3 months prior to dosing.
* Hospitalization due to liver disease within the preceding 1 month prior to dosing.
* Participant has received liver transplant at any time in the past and is on immunosuppressant therapy.
* Participants requiring paracentesis more than every 3 weeks for the management of ascites are excluded.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-06 (Estimated); Primary Completion 2025-06-26 (Estimated); Study Completion 2025-06-26 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-versus-time curve (AUC) from time zero to the last measurable plasma concentration (AUClast) of TNO155 | Up to 240 hours post single dose
  AUClast will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
AUC from time zero to time "t" (AUC0-t) of TNO155 | Up to 240 hours post single dose
  AUC0-t will be calculated as needed based on TNO155 plasma concentrations and non-compartmental methods. The definition of time "t" may be data-driven post-hoc to mitigate treatment bias due to within participant differences in Tlast between the treatments, or may be selected to allow between-study exposure comparisons that use a common time window.
AUC from time zero to infinity (AUCinf) of TNO155 | Up to 240 hours post single dose
  AUCinf will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Maximum (peak) observed plasma concentration (Cmax) of TNO155 | Up to 240 hours post single dose
  Cmax will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Time to reach maximum observed plasma concentration (Tmax) of TNO155 | Up to 240 hours post single dose
  Tmax will be calculated based on TNO155 plasma concentrations and non-compartmental methods
Elimination half-life (T1/2) of TNO155 | Up to 240 hours post single dose
  T1/2 will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Sampling time of the last measurable plasma concentration (Tlast) of TNO155 | Up to 240 hours post single dose
  Tlast will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Apparent plasma clearance (CL/F) of TNO155 | Up to 240 hours post single dose
  CL/F will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Apparent volume of distribution during terminal phase (Vz/F) of TNO155 | Up to 240 hours post single dose
  Vz/F will be calculated based on TNO155 plasma concentrations and non-compartmental methods.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days post single dose
  Incidence of AEs and SAEs, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.
Unbound Cmax (Cmax,u) of TNO155 | Up to 240 hours post single dose
  Cmax,u will be calculated based on the unbound fraction of TNO155 in plasma.
Unbound AUClast (AUClast,u) of TNO155 | Up to 240 hours post single dose
  AUClast,u will be calculated based on the unbound fraction of TNO155 in plasma.
Unbound AUCinf (AUCinf,u) of TNO155 | Up to 240 hours post single dose
  AUCinf,u will be calculated based on the unbound fraction of TNO155 in plasma
Unbound CL/F (CL/F,u) of TNO155 | Up to 240 hours post single dose
  CL/F,u will be calculated based on the unbound fraction of TNO155 in plasma.
Renal clearance (CLr) of TNO155 | Up to 240 hours post single dose
  CLr will be calculated based on urinary excretion data of TNO155.
Apparent non-renal clearance (CLNR/F) of TNO155 | Up to 240 hours post single dose
  CLNR/F will be calculated based on urinary excretion data of TNO155.
Fraction of dose excreted in urine (fe) of TNO155 | Up to 240 hours post single dose
  Fe will be calculated based on urinary excretion data of TNO155.

IPD SHARING:
Plan to Share IPD: No